CLINICAL TRIAL: NCT02758145
Title: Promotion of Influenza Vaccination in Healthcare Workers During the Recruitment Visit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Service de Médecine Préventive Hospitalière (Other)
Responsible Party: Principal Investigator, Currat Michael, Physician, Service de Médecine Préventive Hospitalière
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MDP-2016-00296-FLU
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Human Influenza Vaccination in Healthcare Workers
MeSH Terms: interventions — Clinical Trials, Phase III as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine information (G1) (Active Comparator): During the recruitment visit at the occupational medicine unit between the 04/29/16 and the 10/31/16, the workers in this group (G1) in addition to their recruitment visit, will benefit from a short intervention given by the nurse concerning the flu, the advantages of the flu vaccination, and how they can be vaccinated in the institution. The nurse also transmits an information sheet concerning the benefits of the vaccination. 2 weeks after the beginning of the next flu vaccination campaign, they will receive a reminder letter to encourage vaccination.
  Interventions: Other: Flu vaccination information in 3 phases
- No information (G2) (No Intervention): Workers in the control group (G2) receive no intervention, only recruitment visit.

INTERVENTIONS:
Other: Flu vaccination information in 3 phases — An oral information is given by the nurse during the recruitment visit at the occupational medicine unit. She initiates the discussion on flu and asks the employee if he usually receives the vaccine. Then she provides a brief standardized information on recommendations concerning flu vaccination, and the annual influenza vaccination campaign in CHUV and PMU. She responds to questions.
  After the interview, she gives an informative document with key messages (information about the disease, benefits to be vaccinated, vaccine safety, etc.). The document includes frequently asked questions, website address, and the email address of the occupational medicine unit in case of questions.
  The third phase consists of sending to the employee shortly after the start of the next campaign of flu vaccination (November 2016), a postal mail recalling the information provided during the recruitment examination and inviting them to get vaccinated.
  Arms: Influenza vaccine information (G1)

SUMMARY:
The investigators will compare two groups, an intervention group with a control group. Each employee of the University Hospital of Lausanne (CHUV) and the University Medical Policlinic of Lausanne (PMU) who will do his recruitment visit at the occupational medicine unit of the CHUV between 04/29/16 (end of previous influenza epidemic) and 31/10/16 (the day before the start of the next influenza vaccination campaign) and exert a function in regular contact with patients will be eligible. Depending on his employee number (assigned by the human resources administration, independent of any parameter), he will be placed in the intervention group G1 (odd number) or in the control group G2 (even number). The information concerning the distribution of these two groups will be noted in the computerized medical records of the employee at the occupational medicine unit (Medipho4D software, secured database). Thereafter, the employee will be received by the nurse of the he occupational medicine unit for a recruitment visit according to the usual process. The nurse will perform the study intervention in addition to the usual procedure if it is stipulated ''intervention group'' on the employee's record in the database or only perform the usual steps if it is stipulated ''control group''. At the beginning of the next influenza vaccination campaign (mid-November 2016), employees in the intervention group will receive a letter reminding then about the intervention given during the recruitment visit and inviting them to get vaccinated. During the next influenza vaccination campaign (11.01.16) and until the end of the influenza epidemic that will follow (April 2017), each employee will have the opportunity to be vaccinated at the different vaccination stalls set up by the occupational medicine unit. For each employee vaccinated, the date of vaccination and vaccine name is entered in the electronic medical records of the occupational medicine unit (Medipho4D software) by a nurse or a secretary of the unit. At the end of the human influenza epidemic (April 2017), the data will be extracted from the database (Medipho4D software) and anonymized by an individual not implicated in the study. Data from two groups will be analyzed and compared to assess whether the intervention conducted among newly hired employees promotes influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Employees of CHUV (University Hospital of Lausanne) or PMU (University Policlinic of Lausanne) who work regularly in contact with patients
* Employees who must do the recruitment visit at the occupational medicine unit of the CHUV

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination rate | one year

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Currat M, Lazor-Blanchet C, Zanetti G. Promotion of the influenza vaccination to hospital staff during pre-employment health check: a prospective, randomised, controlled trial. J Occup Med Toxicol. 2020 Nov 18;15(1):34. doi: 10.1186/s12995-020-00285-w. PMID 33292400